CLINICAL TRIAL: NCT05033522
Title: Phase II/III Randomized, Controlled Clinical Study of AlloStim(R) vs Physician's Choice in Asian Subjects With Advanced Hepatocellular Carcinoma
Brief Title: Immunotherapy for Advanced Liver Cancer
Acronym: ALIVE
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor unable to fund
Sponsor: Mirror Biologics, Inc. (Industry)
Collaborators: Immunovative (Thailand) Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBI-003-LIVE
Record Dates: First submitted 2021-08-25; First posted 2021-09-02 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; immunotherapy; Thailand; Malaysia
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Folfox protocol; Sorafenib; lenvatinib

STUDY DESIGN:
Intervention Model Description: Subjects are randomized 2:1 to experimental vs physician's choice. A two-sided logrank test with an overall sample size of 130 subjects (43 in the control group and 87 in the treatment group) achieves 80% power to detect at a 0.05 significance level a hazard ratio of 0.56 when the control group median survival is 6.5 months. A total of 150 subjects are planned to be accrued.
Who Masked: Outcomes Assessor
Masking Description: The investigator and subjects will be informed of the treatment group to which the subject has been randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AlloStim® (Experimental): AlloStim® is a formulation of living allogeneic Th1-like cells with anti-CD3/CD28 microbeads attached derived from precursors purified from healthy screened blood donors that are differentiated and expanded ex-vivo. AlloStim® is formulated at 10-7 cells/ml in 0.5ml for ID administration and 3ml for IV administration
  Interventions: Biological: AlloStim® immunotherapy
- Physician's Choice (Active Comparator): Physician's Choice is sorafenib or levantinib or FOLFOX4 monotherapy
  Interventions: Drug: FOLFOX regimen; Drug: Sorafenib; Drug: Lenvatinib

INTERVENTIONS:
Biological: AlloStim® immunotherapy — 3 cycles of intradermal and intravenous administrations
  Arms: AlloStim®
Drug: FOLFOX regimen — Comparative arm: Physician Choice of FOLFOX4 chemotherapy
  Other Names: Physician Choice FOLFOX4
  Arms: Physician's Choice
Drug: Sorafenib — Comparative arm: Physician Choice of Sorafenib
  Other Names: Sorafenib Physician's Choice
  Arms: Physician's Choice
Drug: Lenvatinib — Comparative Arm: Physician's Choice of Levantinib
  Other Names: Levantinib Physician's Choice
  Arms: Physician's Choice

SUMMARY:
This is a randomized, controlled multi-site, multi-national clinical trial conducted in Thailand and Malaysia for Asian adults (males or females), 18 years of age and older presenting with advanced HCC (BCLC stage C) including subjects with macrovascular involvement and/or extrahepatic spread (not eligible for TACE, surgery or locoregional treatment) with Child-Pugh stage A or B liver function. 150 subjects will be randomized 2:1 to AlloStim® immunotherapy vs Physician's Choice of Sorafenib, Lenvatinib or FOLFOX4.

DETAILED DESCRIPTION:
A multi-national, randomized, controlled trial (RCT) with multiple sites selected in Asia (Malaysia and Thailand). Subjects with no prior treatments for BCLC stage C disease and presenting with Child-Pugh class A or B liver reserve to be randomized 2:1 to AlloStim® vs. Physician's Choice (PC). PC to be declared prior to randomization. PC allowed to be either sorafenib, levantinib or FOLFOX4.

The world incidence of hepatocellular carcinoma (HCC) is highest in East and South East Asia, with nearly half of the all HCC cases and deaths globally occurring in China. In Asian countries, the main treatment options for early or intermediate HCC (BCLC class A and B) include surgical resection, ablation (e.g., RFA, ETOH, cryoablation), transarterial chemoembolization (TACE), radiation or systemic chemotherapy depending on liver function status. However, in the Asian-Pacific region it is estimated that up to 80% of patients present with unresectable, advanced HCC (BCLC Stage C) that are not eligible for locoregional therapy, surgery or TACE due to tumor size and/or vascular involvement. For these patients, the standard of care for over a decade has been sorafenib (Bayer, A.G.), a oral kinase inhibitor based on the results of a RCT (SHARP study) of 602 patients randomized to sorafenib vs. placebo. Median overall survival (OS) was 10.7 months for sorafenib and 7.9 months for placebo (p<0.05). The SHARP study included a Western population. A separate study in Asian patients (226 patients from China, South Korea and Taiwan) comparing sorafenib to placebo (Sorafenib-AP study) demonstrated a OS of 6.5 months for sorafenib compared to 4.2 months for placebo (p<0.05). The placebo OS difference between Asian and Western patients (4.2mo vs 7.9 mo) suggests a difference in the disease characteristics in the Asian population. One significant difference is that the Asian population has an increased prevalence of HBV compared to Western population which may contribute to the increased incidence of HCC and worse OS outcomes observed in Asian patients compared to Western patients.

In Thailand and Malaysia sorafenib is not available to a majority of the population presenting with advanced HCC, both due to cost and toxicity profile. This study is designed to evaluate whether AlloStim ® immunotherapy will provide a survival benefit to this population with an improved quality of life compared to approved first line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who are at least 18 years of age at time of enrollment
2. Histologically or cytologically documented advanced HCC (BCLC stage C) disease at diagnosis.
3. No prior treatment for BCLC class C disease.
4. Child-Pugh Class A or subset of Child-Pugh Class B
5. Performance status: ECOG < 2 with no deterioration over the previous 2 weeks
6. With or without positive HBV and/or HCV
7. With or without extrahepatic disease and with or without macrovascular invasion
8. Measurable enhancing disease in liver with at least one target lesion evaluable by mRECIST
9. Adequate hematological, liver and renal function as assessed by the following:

   * Hemoglobin > 10.0 g/dl
   * Platelet count > 75,000/μl
   * ALT and AST < 5.0 x ULN
   * Serum creatinine < 1.5
10. Women of child-bearing potential: negative pregnancy test
11. Patients of child producing potential: usage of contraception or avoidance of pregnancy measures while enrolled on study
12. Ability to understand the study, its inherent risks, side effects and potential benefits and ability to give written informed consent to participate

Exclusion Criteria:

1. Any prior cancer diagnosis (other than cured basal cell carcinoma, head and neck carcinoma in-situ, or superficial Ta, Tis, T1 bladder cancer) or concurrent cancer histologically different than HCC (e.g., cholangiocarcinoma).
2. Child-Pugh liver function combined score >9 (Class C or Class D)
3. Moderate uncontrolled or severe ascites (+3 on Child-Pugh calculator)
4. Clinical symptoms of hepatic decompensation or presence of hepatic encephalopathy
5. Severe stomach/esophageal varices requiring interventional treatment.
6. Unable to tolerate radiological contrast dye
7. Any prior experimental, approved or off-label treatment for HCC (including levantinib, nivolumab, duvalumab, tremelimumab, brivananib, cabozantinib or ramucircumab) or any approved or experimental procedures such as surgery, radiation or ablation.
8. Enrollment in any previous clinical trial for HCC
9. Any history of autoimmune disorder (type I, insulin-dependent diabetes allowed)
10. History of COPD or oxygen saturation <92% at room air
11. Any clinical condition requiring systemic steroids (inhaled steroids allowed) or any current immunosuppressive therapy or anti-epileptic drug therapy.
12. Known history of HIV infection
13. Clinically significant gastrointestinal bleeding within 30 days prior to study entry
14. History of cardiac disease: congestive heart failure > NYHA class 2; cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or Digoxin are permitted)
15. Uncontrolled hypertension (SBP >150 or DBP>90).
16. Active clinically serious infections (> grade 2 CTCAE version 5.0)
17. History of organ transplant or tissue allograft
18. Uncontrolled concurrent serious medical or psychiatric illness
19. Clinically apparent central nervous system metastases or carcinomatous meningitis
20. History of drug abuse or current alcohol abuse
21. History of blood transfusion reactions
22. Pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | rom date of randomization until the date of death from any cause, assessed up to 48 months
  the time from randomization till death

SECONDARY OUTCOMES:
Quality of Life Survey | weekly assessments from baseline to 28 weeks
  using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) and the Functional Assessment of Cancer Therapy-Hepatobiliary Questionnaire (FACT-Hep)
Time to Symptomatic Progression | rom date of randomization weekly for up to 24 weeks until the date of first documented progression which ever comes first
  To assess time to symptomatic progression (TTSP)

CONTACTS AND LOCATIONS:
Locations (8):
- Malaysia (3):
  - Sultan Ismail Hospital, Johor Bahru, Johor
  - Sultanah Bahiyah Hospital, Alor Star, Kedah
  - Columbia Asia Bukit Rimau, Shah Alam, Selangor
- Thailand (5):
  - Siriraj Hospital, Bangkok Noi, Bangkok
  - Prince of Songkla University (Songklanagarind Hospital), Hat Yai, Changwat Songkhla
  - Naresuan University Hospital, Phitsanulok, Tha Pho
  - Chiangmai University, Chiang Mai
  - Songklanagarind Hospital, Khon Kaen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: sponsor website — http://www.mirrorbio.com